CLINICAL TRIAL: NCT02624362
Title: The Effect of Suggestion of Harmful/Beneficial Effects of Odors on Asthma Symptoms
Brief Title: The Effect of Odors on Asthma Symptoms
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Collaborators: KU Leuven (Other); Research Foundation Flanders (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: S57940
Record Dates: First submitted 2015-12-01; First posted 2015-12-08 (Estimated); Last update posted 2024-07-03 (Actual); Status verified 2024-07

CONDITIONS: Asthma
Keywords: Odor; trigger; inflammation; nocebo
MeSH Terms: conditions — Asthma; Inflammation | interventions — Suggestion; Ethanol; Odorants

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Odor+ Positive belief (Experimental): Participants receive 15 minute odor presentation (Phenylethyl Alcohol odor) accompanied by the suggestion that this odor improves asthma symptoms (therapeutic suggestion)
  Interventions: Behavioral: Therapeutic Suggestion; Other: Phenylethyl Alcohol odor
- Odor + Negative belief (Experimental): Participants receive 15 minute odor presentation (Phenylethyl Alcohol odor) accompanied by the suggestion that this odor worsens asthma symptoms (asthmogenic suggestion)
  Interventions: Behavioral: Asthmogenic Suggestion; Other: Phenylethyl Alcohol odor

INTERVENTIONS:
Behavioral: Therapeutic Suggestion — suggestions about potential beneficial effects of the odor are given
  Other Names: placebo suggestion; positive treatment belief induction
  Arms: Odor+ Positive belief
Behavioral: Asthmogenic Suggestion — suggestions about potential negative effects of the odor are given
  Other Names: nocebo suggestion; negative treatment belief
  Arms: Odor + Negative belief
Other: Phenylethyl Alcohol odor — Over the course of 15 minutes, participants, receive 15 short sniffs of Phenylethyl Alcohol odor

SUMMARY:
An extended replication of Jaen & Dalton (2014), the investigators aim to investigate the role of odors and associated trigger beliefs on symptom perception and airway inflammation in individuals with asthma

DETAILED DESCRIPTION:
Participants with asthma are randomly assigned to a 15-min (phenylethyl alcohol) odor inhalation, accompanied by either an asthmogenic suggestion (nocebo), or a therapeutic suggestion (placebo). Airway inflammation, lung function, and asthma symptoms are measured in response to the odor/suggestion, up to 24 hours after odor inhalation. The investigators are also measuring worry and heart rate variability as potential mediators of the response.

ELIGIBILITY:
Inclusion Criteria:

* A physician diagnosis of asthma

Exclusion Criteria:

* FEV1 lower than 60% predicted
* clinical condition other than asthma

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2015-08 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline Exhaled Nitric Oxide to 24 hours after odor induction | baseline, immediately after odor induction, 2 hours after odor induction, 24 hours after odor induction
  Fraction of exhaled nitric oxide

SECONDARY OUTCOMES:
asthma symptoms | baseline, immediately after odor induction, 2 hours after odor induction, 24 hours after odor induction
  measured using the Asthma Symptom Checklist
Forced Expiratory Volume at one second (FEV1) | baseline, immediately after odor induction, 2 hours after odor induction, 24 hours after odor induction
  Measured using Jaeger Masterscreen Spirometer, according to ERS-ATS guidelines
Worry | baseline, immediately after odor induction, 2 hours after odor induction, 24 hours after odor induction
  measured using worry Visual Analog Scales
Cortisol | baseline, immediately after odor induction, 2 hours after odor induction, at awakening, 30 min after awakening, 24 hours after odor induction
  cortisol awakening response (AUC), and changes in cortisol (AUC) will be measured using saliva sampling
Change in Heart rate and Heart Rate Variability (HRV) | change from baseline to 24 hours after odor induction
  24 hour heart rate data will be recorded using an ambulatory ECG monitor, and analyzed in 1 hour epochs, extracting mean of successive differences (MSD) as a variable of interest.
Change in Respiratory rate | change from baseline to 15 min odor presentation
  respiratory rate (breaths/min) is recorded continuously, and changes between baseline and odor presentation periods will be analysed
change in Fraction of end-tidal carbon dioxide (FetCO2) | change from baseline to 15 min odor presentation
  FetCO2 (plateau %CO2 in exhaled air) is recorded continuously, and changes between baseline and odor presentation periods will be analysed

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Janssens, PhD, Principal Investigator — KU Leuven
Locations (1):
- UZ Leuven, Leuven, Belgium